CLINICAL TRIAL: NCT02721784
Title: Serial mpMRI (Multi Parametric Magnetic Resonance Imaging) Scanning in Prostate Cancer After Androgen Deprivation Therapy and RadioTherapy (SMART)
Brief Title: Serial mpMRI (Multi Parametric Magnetic Resonance Imaging) Scanning in Prostate Cancer After Androgen Deprivation Therapy and RadioTherapy
Acronym: SMART
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15/0342
Record Dates: First submitted 2016-01-04; First posted 2016-03-29 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
Keywords: MRI; Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pre- and Post- Radiotherapy MRI (Other): mpMRI/VERDICT sequences to be preformed pre- and post- EBRT (external beam radiotherapy) according to the following schedule:
  Pre-Androgen Deprivation Therapy 3 weeks before radiotherapy 6 week after starting radiotherapy 6 Months after starting radiotherapy
  External Beam Radiotherapy to be given after 3 months of androgen deprivation
  Interventions: Device: mpMRI/VERDICT; Radiation: External Beam Radiotherapy

INTERVENTIONS:
Device: mpMRI/VERDICT — Combined MRI sequences of T2, DCE, Diffusion and VERDICT
Radiation: External Beam Radiotherapy — 78Gy (Gray) to Prostate +/- Pelvic

SUMMARY:
The evaluation of the radiological changes in localised or locally advanced prostate cancer after androgen deprivation therapy and external beam radiotherapy using multi-parametric MRI (multi parametric magnetic resonance imaging) and VERDICT (Vascular, Extracellular and Restricted Diffusion for Cytometry in Tumours) sequences.

DETAILED DESCRIPTION:
External beam radiotherapy (EBRT) fails to eradicate prostate cancer in 24-33% of cases. Response is monitored solely by testing serum prostate specific antigen (PSA), with biochemical failure following radiotherapy defined as a prostate specific antigen (PSA) level of 2 ng/ml above the nadir.

T2 and Dynamic Contrast Enhanced (DCE) MRI have been shown to be able to detect the recurrence of prostate cancer following radiotherapy. Changes seen in Apparent Diffusion Coefficient (ADC) variables post-treatment have potential use in monitoring disease response to radiotherapy but the natural history of these changes during and after treatment remains uncertain and warrants further investigation.

This study investigates the feasibility of using multi-parametric MRI (mpMRI) and novel diffusion-weighted sequences called VERDICT (Vascular, Extracellular and Restricted Diffusion for Cytometry in Tumours) at various stages during the treatment of prostate cancer with radiotherapy. Patients will be first scanned before androgen deprivation therapy (ADT) starts, then 3 weeks before the start of radiotherapy, again in week 6 of radiotherapy and once more 6 months after the end of radiotherapy. In addition, all patients entered into the study will already have had a mpMRI scan prior to prostate biopsy as part of their standard care.

Multi-parametric MRI and VERDICT sequences may reveal changes in the tumour and normal prostate before a detectable PSA increase. This could allow for their use in response assessment following radiotherapy and androgen deprivation treatment. If such clinical utility is proven, referral for salvage treatment using High Intensity Focussed Ultrasound (HIFU), cryotherapy or salvage radical prostatectomy may be expedited.

ELIGIBILITY:
Inclusion Criteria:

1. Targeted or Concordant biopsy confirmed prostate cancer
2. Pre-biopsy mpMRI scan of the prostate undertaken at University College London Hospital (UCLH)
3. Agrees to have ADT and EBRT

Exclusion Criteria:

1. Treatment within the previous 6 months with any form of hormones (including 5-alpha reductase inhibitors)
2. Evidence of metastatic disease
3. Prior local intervention to the prostate
4. Unable to give informed consent
5. Any prosthesis (including hip replacements) which could cause artefacts degrading the quality of the imaging
6. Contraindication to gadolinium contrast agent
7. Unable to tolerate an MRI

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of changes in MRI ADC value | 6 months
Measurement of changes in mpMRI tumour volume (cubic centimetres) | 6 months
Measurement of changes in enhancement measured as a transfer constant (KTrans) value | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Research Group, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided